CLINICAL TRIAL: NCT04463888
Title: Development of a Smart Home-based Exoskeleton Robot System and Innovative Service Model for Stroke Patients
Brief Title: A Smart Home-based Exoskeleton Robot System for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B-BR-107-084
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Rehabilitation, Tenodesis, Stroke, Internet of Things
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot training with Smart Home-based Exoskeleton Robot System (Experimental): In addition to receiving hospital occupational therapy training twice a week, the participants will receive 60 minutes of home-based robot assisted tenodesis-grip training per day, 5 days a week, for 4 weeks .
  Interventions: Other: occupational therapy
- control group (Active Comparator): In addition to receiving hospital occupational therapy training twice a week, the participants will receive 60 minutes of home-based specific motor task training per day, 5 days a week, for 4 weeks .
  Interventions: Other: occupational therapy

INTERVENTIONS:
Other: occupational therapy — occupational therapy targeted to goals that are relevant to the functional needs of the patient

SUMMARY:
In the proposed study, the investigators assumed that high dose of repetitive motor task training using an exoskeleton robot-assisted system may provide benefits in motor shaping and greater brain priming for hand paresis of the stroke patients. Nevertheless, the amount of therapeutic activity with clinicians' guidance is often short of number in therapy sessions.Therefore, using Internet of Things (IoT), connected rehabilitation products and the data they generate that are a new trend of rehabilitation strategy for providing remote home-programs support. The specific aim of this study is to to explore the feasibility of introducing the rental services of a Smart Home-based Exoskeleton Robot System through the IoT business model. And the second purpose is to investigate the effects of applying the exoskeleton robotic device for tenodesisgrip training as a home-based treatment for chronic stroke patients.The expected outcomes of this research are to clarify the feasibility of using IoT business model for launching smart rehabilitation device rental service and the effects of application a high dosage of hand movement training as home program on motor and hand function for patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* (1) chronic stroke patients with unilateral cerebral infarction or hemorrhage, (2) computed tomography scan that excluded pathologies other than unilateral cerebral hemisphere injury, (3) capacity to perform a pinch task with the thumb and index finger, (4) no major cognitive or perceptual deficit (i.e., visual, auditory, perceptual, praxis, and memory, as determined using Lowenstein occupational therapy cognitive assessment), (5) premorbid right-handedness and (6) first-ever stroke.

Exclusion Criteria:

* not meeting inclusion criteria, and with Wernicke's aphasia or global aphasia leading to difficulty of following instruction.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the result of Box and blocks test | baseline, 4 weeks, 16 weeks and 20 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change in the result of Fugl-Meyer assessment for UE motor function | baseline, 4 weeks, 16 weeks and 20 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.
Change in the result of Modified Ashworth scale (MAS) | baseline, 4 weeks,16 weeks and 20 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 4 weeks,16 weeks and 20 weeks
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, 4 weeks,16 weeks and 20 weeks
  MAL is a structured interview with testing sensitivity used to examine how much (amount of use, AOU) and how well (quality of movement, QOM) the subject uses their more-affected arm. For the 30 items MAL, each item is scored on a 0-5-ordinal scale.
Clinical global impression scale | post-intervention (week 4)
  Self-reported improvement over the treatment period,. The scale, rated from 1 (very much improved) to 7 (very much worse), is as the indicator for determining perceptible change of the patients for assisted tenodeis-grip robot system.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Kuo LC, Yang KC, Lin YC, Lin YC, Yeh CH, Su FC, Hsu HY. Internet of Things (IoT) Enables Robot-Assisted Therapy as a Home Program for Training Upper Limb Functions in Chronic Stroke: A Randomized Control Crossover Study. Arch Phys Med Rehabil. 2023 Mar;104(3):363-371. doi: 10.1016/j.apmr.2022.08.976. Epub 2022 Sep 16. PMID 36122608